CLINICAL TRIAL: NCT03332927
Title: A Randomized, Crossover Trial to Assess the Effects of Replacing Commonly Consumed Breakfast Foods With Eggs on Insulin Sensitivity and Other Markers of Cardiometabolic Health in Men and Women at Increased Risk for Type 2 Diabetes Mellitus.
Brief Title: Effect of Egg Consumption on Cardiometabolic Health in Prediabetic Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MB-1704
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg based breakfast foods (Experimental): Study products delivering two eggs/day, 6 days per week, will be administered for the 4-week treatment period.
  Interventions: Other: Egg based breakfast foods
- Non-egg based breakfast foods (Active Comparator): Study products delivering non-egg based control breakfast foods will be administered 6 days per week for the 4-week treatment period.
  Interventions: Other: Non-egg based breakfast foods

INTERVENTIONS:
Other: Egg based breakfast foods — Two eggs/day, 6 days per week provided as breakfast foods such as burrito-type roll-up, egg sandwich and omelet.
  Arms: Egg based breakfast foods
Other: Non-egg based breakfast foods — Non-egg based control foods provided as breakfast foods 6 days per week such as waffles, ready-to-eat cereal, fruits and cheeses.
  Arms: Non-egg based breakfast foods

SUMMARY:
The objective of this trial is to assess the effects of whole egg consumption (12 per week), compared to energy-matched typical breakfast control foods, on insulin sensitivity and other markers of metabolic health, including fasting lipoprotein lipid levels and resting blood pressure.

DETAILED DESCRIPTION:
This is a randomized, crossover study that includes two screening visits and two 4-week test periods separated by a 4-week washout. Subjects will consume two eggs/day (12 eggs/week consumed over 6 days per week, provided as breakfast foods such as burrito-type roll-up, egg sandwich and omelet) or non-egg based control foods (provided as breakfast foods such as English muffins, bagels, ready-to-eat cereal, and flavored muffins). The background diet will be a habitual diet. The nutritional profiles of the egg and control breakfast foods will be designed such that the energy from eggs will be substituted for a mixture of carbohydrate, protein and fat in the control foods.

Study foods will be dispensed with instructions to consume the assigned breakfast food starting on day 1. Subjects will be instructed to consume the breakfast foods in their entirety each day, for the duration of the 28 day test period, and to record daily study food intake. Subjects will receive diet instruction on the incorporation of food substitutions during the test period to maintain habitual energy intake. Compliance will be assessed using the Daily Log intake and number of foods consumed based on returned foods.

An intravenous glucose tolerance test (IVGTT) will be completed at baseline and the end of each treatment period for evaluation of insulin sensitivity. Blood will be collected for a fasting lipid profile (at all visits), glucose and insulin, high-sensitivity C-reactive protein (hs-CRP), vertical auto profile (VAP) for cholesterol carried by lipoprotein fractions (at baseline and end of each treatment period), with additional blood samples collected for storage and archived for possible future analysis of non-genetic indicators of metabolism. Assessments of vital signs and body weight, review of concomitant medication/supplement use and inclusion and exclusion criteria for relevant changes, and evaluation of adverse effects will be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of ≥25.0 kg/m2 (≥23.0 kg/m2 in Asian Americans) to 39.99 kg/m2.
2. Metabolic syndrome [exhibiting at least 3 out of 5 of these criteria]: waist circumference ≥102 cm (40 inches) in men or ≥88 cm (35 inches) in women, TG level ≥150 mg/dL, HDL-C level <40 mg/dL in men or <50 mg/dL in women, hypertension: ≥130 systolic and/or /≥85 diastolic or on drug therapy for elevated BP, fasting hyperglycemia: 100-125 mg/dL.
3. Prediabetes [exhibiting any of the criteria below at screening]: glycated hemoglobin 5.7-6.4% (inclusive), or fasting capillary glucose of 100-125 mg/dL (inclusive), or a 2-h postprandial glucose of 140-199 mg/dL.

Exclusion Criteria:

1. Atherosclerotic cardiovascular disease including any of the following:

   clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., myocardial infarction, angina, transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound] or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
2. History or presence of clinically important pulmonary (including uncontrolled asthma), endocrine (including type 1 or 2 diabetes mellitus), chronic inflammatory disease (including irritable bowel disease, lupus, rheumatoid arthritis), hepatic, renal, hematologic, immunologic, neurologic, or biliary disorders.
3. Known allergy, sensitivity, or intolerance to any ingredients in the study foods.
4. Uncontrolled hypertension
5. Recent history of cancer in the prior 5 years, except for non-melanoma skin cancer.
6. Recent change in body weight of ±4.5 kg.
7. Unstable use of any antihypertensive medication.
8. Recent use of any medications intended to alter the lipid profile [e.g. bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin (drug form), omega-3-ethyl ester drugs, and/or proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitors], weight-loss drugs, systemic corticosteroid drugs, medications known to influence carbohydrate (CHO) metabolism [e.g. adrenergic receptor blockers, thiazide diuretics, hypoglycemic medications], and/or anti-psychotics.
9. Recent use of foods or dietary supplements that might influence lipid metabolism [e.g. omega-3 fatty acid supplements (e.g., fish or algal oils) or fortified foods, sterol/stanol products; dietary supplements (red rice yeast supplements; garlic supplements; soy isoflavone supplements; niacin or its analogues at doses >400 mg/d], inconsistent use of Metamucil® or viscous fiber-containing supplements
10. Use of antibiotics within 5 days of screening.
11. Pregnant, planning to be pregnant during the study period, lactating, or of childbearing potential and unwilling to commit to the use of a medically approved form of contraception throughout the study period.
12. Extreme dietary habits (e.g., vegan or very low carbohydrate diet).
13. Current or recent history or strong potential, for drug or alcohol abuse.
14. History of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
15. Recent exposure to any non-registered drug product.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity index (IV-SI) from short (40 min) IVGTT. | Up to 40 minutes - measured at baseline and end of each treatment period.
  Percent change or change from baseline to end of each treatment condition

SECONDARY OUTCOMES:
Disposition index [acute insulin response to intravenous glucose (AIRg) x IV-SI] | Up to 40 minutes - measured at baseline and end of each treatment period.
  Percent change (or change) from baseline to the end of each treatment period.
Glucose fractional disappearance rate from t = 10-40 min (Kg) | Up to 40 minutes - measured at baseline and end of each treatment period.
  Percent change (or change) from baseline to the end of each treatment period.
Homeostasis model assessments of insulin sensitivity (HOMA%S) | Up to 29 days for each treatment period
  Percent change (or change) from baseline to the end of each treatment period.
Beta-cell function (HOMA%B) | Up to 29 days for each treatment period
  Percent change (or change) from baseline to the end of each treatment period.
Percent change in Total cholesterol (TC) | Up to 29 days for each treatment period
  Percent change in TC from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Percent change in low-density lipoprotein cholesterol (LDL-C) | Up to 29 days for each treatment period
  Percent change in LDL-C from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Percent change in high-density lipoprotein cholesterol (HDL-C) | Up to 29 days for each treatment period
  Percent change in HDL-C from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Percent change in non-HDL-C | Up to 29 days for each treatment period
  Percent change in non-HDL-C from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Percent change in TC/HDL-C ratio | Up to 29 days for each treatment period
  Percent change in TC/HDL-C ratio from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Percent change in Triglycerides (TG) | Up to 29 days for each treatment period
  Percent change in TG from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Seated, resting systolic and diastolic blood pressure (BP) | Up to 29 days for each treatment period
  Percent change in seated, resting systolic and diastolic BP (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)
Vertical Auto-Profile (VAP) analysis of cholesterol carried by lipoproteins and lipoprotein subfractions. | Up to 29 days for each treatment period
  Percent change in VAP analysed cholesterol in lipoproteins and lipoprotein subfractions from baseline (average of the values from one screening visit and the baseline visit) to the end of each test condition (average of the values at 3-week and 4-week visits of each test period)

CONTACTS AND LOCATIONS:
Locations (1):
- Great Lakes Clinical Trials, Chicago, Illinois, United States